CLINICAL TRIAL: NCT01024803
Title: Safety and Efficacy of Subretinal Implants for Partial Restoration of Vision in Blind Patients: A Prospective Multicenter Clinical Study Based on Randomized Intra-individual Implant Activation in Patients With Degenerative Retinal Diseases
Brief Title: Safety and Efficacy of Subretinal Implants for Partial Restoration of Vision in Blind Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Implant AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RI-MC-CT-2009
Record Dates: First submitted 2009-11-26; First posted 2009-12-03 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Retinitis Pigmentosa; Retinal Degeneration
Keywords: Retina implant, Subretinal; Legal blindness; Genetic Diseases, Inborn; Eye Diseases; Retinitis Pigmentosa; Retinitis; Retinal Degeneration; Eye Diseases, Hereditary; Retinal Diseases
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Degeneration; Blindness; Genetic Diseases, Inborn; Eye Diseases; Retinitis; Eye Diseases, Hereditary; Retinal Diseases | interventions — Visual Prosthesis; Eye, Artificial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Device name: "Retina Implant model Alpha". Surgical implantation of medical device into eye — Surgical implantation of medical device named "Retina Implant" into eye to restore vision partially.
  Randomized intra-individual implant activation in patient under test conditions such as: FrACT, BaLM, BaGA, maze, ADL.
  Other Names: retinal implant; bionic eye; artificial vision; artificial eye; restoration of vision; eye chip; vision prosthesis; eye implant; retinal prosthesis

SUMMARY:
Patients suffering from hereditary retinal degeneration receive a retinal implant to restore sight.

Subretinal implant "ON" results in significant visual acuity improvement, when compared to "OFF" condition.

ELIGIBILITY:
Inclusion Criteria:

* Hereditary retinal degeneration of the outer retinal layers i.e. photoreceptor rods & cones.
* Pseudophakia
* Angiography shows retinal vessels adequately perfused, despite pathological RP condition.
* Age between 18 and 78 years.
* Blindness (at least monocular) i.e. visual functions not appropriate for localization of objects, self sustained navigation and orientation.
* Ability to read normal print in earlier life, optically corrected without magnifying glass.
* Willing and able to give written informed consent in accordance to EN ISO 14155 (section 6.7) and local legislation prior to participation in the study. Able to perform the study during the full time period of one year for Module-2.

Exclusion Criteria:

* Period of appropriate visual functions approx. 12 years / lifetime.
* Optical Coherence Tomography (OCT) shows significant retina edema &/or scar tissue within target region for implant.
* Retina detected as too thin to expect required rest-functionality of inner retina as shown via Optical Coherence Tomography (OCT).
* Lack of inner-retinal function, as determined by Electrically Evoked Phosphenes (EEP).
* Heavy clumped pigmentation at posterior pole
* Any other ophthalmologic disease with relevant effect upon visual function (e.g. glaucoma, optic neuropathies, trauma, diabetic retinopathy, retinal detachment).
* Amblyopia reported earlier in life on eye to be implanted
* Systemic diseases that might imply considerable risks with regard to the surgical interventions and anaesthesia (e.g. cardiovascular/ pulmonary diseases, severe metabolic diseases).
* Neurological and/or psychiatric diseases (e.g. M. Parkinson, epilepsy, depression).
* Hyperthyroidism or hypersensitivity to iodine
* Women who are pregnant or nursing, or women of childbearing potential who are not willing to use a medically acceptable means of birth control for the duration of the study, or women unwilling to perform a pregnancy test before entering the study.
* Participation in another interventional clinical trial within the past 30 days.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-12; Primary Completion 2017-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Activities of daily living and mobility significantly improve with implant-ON shown via activities of daily living tasks, recognition tasks, mobility, or a combination thereof. | every 3 months for a period of one year

SECONDARY OUTCOMES:
Visual acuity/light-perception and/or object-recognition are significantly improved with implant-ON versus OFF as shown via: FrACT/BaLM/BaGA/VFQ-25 or a combination thereof. | every 3 months for a period of one year
Patient long term safety and stability of implant function | every 3 months for a period of one year

CONTACTS AND LOCATIONS:
Overall Officials: Eberhart Zrenner, Prof. MD, Study Chair — Centre for Ophthalmology, Institute for Ophthalmic Research, University of Tuebingen, Germany; Karl-Ulrich Bartz-Schmidt, Prof. MD, Principal Investigator — University Eye Hospital Tuebingen, Germany; Timothy L Jackson, PhD FRCOphth, Principal Investigator — King's College Hospital NHS Trust; János Németh, Prof. MD PhD, Principal Investigator — Department of Ophthalmology Semmelweis University Budapest; Robert E MacLaren, Prof. DPhil, Principal Investigator — Department of Ophthalmology, John Radcliffe Hospital, Oxford, UK; Johann Roider, Prof. MD, Principal Investigator — University Eye Hospital, Kiel, Germany; Helmut Sachs, PD, MD, Principal Investigator — Eye Hospital Dresden-Friedrichstadt, Germany
Locations (6):
- Germany (3):
  - Helmut Sachs, MD, PD, Dresden
  - Johann Roider, MD, Prof., Kiel
  - Karl-Ulrich Bartz-Schmidt, MD, Prof., Tübingen
- Miklos Resch, MD, PhD, Budapest, Hungary
- United Kingdom (2):
  - Timothy L Jackson, MB.ChB, PhD, FRCOphth, London
  - Robert MacLaren, MD, Prof., DPhil DipEd FRCOphth FRCS, Oxford

REFERENCES:
- [Background] Koitschev A, Stingl K, Bartz-Schmidt KU, Braun A, Gekeler F, Greppmaier U, Sachs H, Peters T, Wilhelm B, Zrenner E, Besch D. Extraocular Surgical Approach for Placement of Subretinal Implants in Blind Patients: Lessons from Cochlear-Implants. J Ophthalmol. 2015;2015:842518. doi: 10.1155/2015/842518. Epub 2015 Dec 10. PMID 26783453
- [Background] Hafed ZM, Stingl K, Bartz-Schmidt KU, Gekeler F, Zrenner E. Oculomotor behavior of blind patients seeing with a subretinal visual implant. Vision Res. 2016 Jan;118:119-31. doi: 10.1016/j.visres.2015.04.006. Epub 2015 Apr 20. PMID 25906684
- [Background] Stingl K, Gekeler F, Bartz-Schmidt KU, Kogel A, Zrenner E, Gelisken F. Fluorescein angiographic findings in eyes of patients with a subretinal electronic implant. Curr Eye Res. 2013 May;38(5):588-96. doi: 10.3109/02713683.2013.767349. Epub 2013 Feb 14. PMID 23410193
- [Background] Stingl K, Bartz-Schmidt KU, Besch D, Braun A, Bruckmann A, Gekeler F, Greppmaier U, Hipp S, Hortdorfer G, Kernstock C, Koitschev A, Kusnyerik A, Sachs H, Schatz A, Stingl KT, Peters T, Wilhelm B, Zrenner E. Artificial vision with wirelessly powered subretinal electronic implant alpha-IMS. Proc Biol Sci. 2013 Feb 20;280(1757):20130077. doi: 10.1098/rspb.2013.0077. Print 2013 Apr 22. PMID 23427175
- [Result] Stingl K, Bartz-Schmidt KU, Besch D, Chee CK, Cottriall CL, Gekeler F, Groppe M, Jackson TL, MacLaren RE, Koitschev A, Kusnyerik A, Neffendorf J, Nemeth J, Naeem MA, Peters T, Ramsden JD, Sachs H, Simpson A, Singh MS, Wilhelm B, Wong D, Zrenner E. Subretinal Visual Implant Alpha IMS--Clinical trial interim report. Vision Res. 2015 Jun;111(Pt B):149-60. doi: 10.1016/j.visres.2015.03.001. Epub 2015 Mar 23. PMID 25812924
- [Result] Kitiratschky VB, Stingl K, Wilhelm B, Peters T, Besch D, Sachs H, Gekeler F, Bartz-Schmidt KU, Zrenner E. Safety evaluation of "retina implant alpha IMS"--a prospective clinical trial. Graefes Arch Clin Exp Ophthalmol. 2015 Mar;253(3):381-7. doi: 10.1007/s00417-014-2797-x. Epub 2014 Sep 16. PMID 25219982
- [Result] Stingl K, Bartz-Schmidt KU, Gekeler F, Kusnyerik A, Sachs H, Zrenner E. Functional outcome in subretinal electronic implants depends on foveal eccentricity. Invest Ophthalmol Vis Sci. 2013 Nov 19;54(12):7658-65. doi: 10.1167/iovs.13-12835. PMID 24150759
- [Result] Stingl K, Schippert R, Bartz-Schmidt KU, Besch D, Cottriall CL, Edwards TL, Gekeler F, Greppmaier U, Kiel K, Koitschev A, Kuhlewein L, MacLaren RE, Ramsden JD, Roider J, Rothermel A, Sachs H, Schroder GS, Tode J, Troelenberg N, Zrenner E. Interim Results of a Multicenter Trial with the New Electronic Subretinal Implant Alpha AMS in 15 Patients Blind from Inherited Retinal Degenerations. Front Neurosci. 2017 Aug 23;11:445. doi: 10.3389/fnins.2017.00445. eCollection 2017. PMID 28878616
- [Derived] Cehajic Kapetanovic J, Troelenberg N, Edwards TL, Xue K, Ramsden JD, Stett A, Zrenner E, MacLaren RE. Highest reported visual acuity after electronic retinal implantation. Acta Ophthalmol. 2020 Nov;98(7):736-740. doi: 10.1111/aos.14443. Epub 2020 Apr 28. PMID 32343050
- [Derived] Kuehlewein L, Troelenberg N, Stingl K, Schleehauf S, Kusnyerik A, Jackson TL, MacLaren RE, Chee C, Roider J, Wilhelm B, Gekeler F, Bartz-Schmidt KU, Zrenner E, Stingl K. Changes in microchip position after implantation of a subretinal vision prosthesis in humans. Acta Ophthalmol. 2019 Sep;97(6):e871-e876. doi: 10.1111/aos.14077. Epub 2019 Feb 28. PMID 30816625
- [Derived] Rock T, Bartz-Schmidt KU, Bramkamp M, Rock D. Influence of axial length on thickness measurements using spectral-domain optical coherence tomography. Invest Ophthalmol Vis Sci. 2014 Oct 8;55(11):7494-8. doi: 10.1167/iovs.14-14043. PMID 25298411
- [Derived] Kusnyerik A, Greppmaier U, Wilke R, Gekeler F, Wilhelm B, Sachs HG, Bartz-Schmidt KU, Klose U, Stingl K, Resch MD, Hekmat A, Bruckmann A, Karacs K, Nemeth J, Suveges I, Zrenner E. Positioning of electronic subretinal implants in blind retinitis pigmentosa patients through multimodal assessment of retinal structures. Invest Ophthalmol Vis Sci. 2012 Jun 20;53(7):3748-55. doi: 10.1167/iovs.11-9409. PMID 22562517